CLINICAL TRIAL: NCT00737815
Title: Magnesium Supplements, Plasma Inflammatory Markers, and Gene Expression in Overweight Individuals With Metabolic Syndrome: a Randomized , Controlled Crossover Trial
Brief Title: Randomized Crossover Study of Magnesium Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Simin Liu, Dr., Director of Genomics and Nutrition, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: GM-LIU; Award No. 200602222; Fund No. 445963-SM-57277
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus, Type 2; Inflammation
Keywords: Randomized Controlled Trial; Magnesium; Diabetes Mellitus, Type 2; Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Inflammation | interventions — Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Magnesium citrate: a total of 500 mg of elemental magnesium
  Interventions: Dietary Supplement: Magnesium Citrate: a total of 500 mg elemental magnesium
- B (Placebo Comparator): Placebo pills
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium Citrate: a total of 500 mg elemental magnesium — 500 mg elemental magnesium
  Arms: A
Other: Placebo — Inactive placebo pill
  Arms: B

SUMMARY:
The investigators recent epidemiologic work in several national surveys and cohorts of men and women have shown that dietary patterns high in plant-based foods and phytochemicals are associated with lower plasma levels of insulin, triglycerides, and C-reactive protein, and reduced risk of type 2 DM and CHD. While the physiologic impact of different foods on serum glucose and insulin is of critical importance, the extent to which specific dietary nutrients can modify insulin resistance is not well understood. Magnesium is a biologically active constituent in whole-grain, green leafy vegetables, and nuts and appears to play an essential role in hundreds of physiologic processes in humans. However, it remains uncertain whether magnesium intake can exert effects on insulin sensitivity and inflammation. Moreover, little is known of the extent to which magnesium intake elicits changes in the expression levels of key genes responsible for glucose homeostasis and systemic inflammation. The ultimate clinical question is whether magnesium supplementation would be clinically effective for the improvement of metabolic disorders in not yet diabetic but high-risk individuals, especially those who are susceptible to insulin resistance. Therefore, as a direct follow up on our previous work in studying the health benefits of plant-based foods such as whole grains, fruits and vegetables, we propose a pilot randomized trial to unravel the metabolic and anti-inflammatory effects of magnesium supplementation versus placebo among overweight individuals with the metabolic syndrome who are particularly prone to the adverse effects of magnesium deficiency. Recent advancements in molecular genetics and genomic technologies have also enabled us to analyze the expression levels of thousands of genes simultaneously in different experimental conditions. The application of high throughput microarray technology in randomized-controlled setting when analyzed with novel statistical methods, will not only help our understanding of nutrient-disease relations, but also afford the investigators the opportunity to gain important insight into the molecular mechanism for complex biological systems of inflammation, insulin resistance, and metabolic abnormalities in response to nutrition intervention.

ELIGIBILITY:
Inclusion Criteria:

* Overweight individuals (with a BMI of ≥ 25 kg/m2)
* Between the ages of 30 and 70 years

Exclusion Criteria:

* Concurrent documented cardiac, or renal disease as recorded by history of myocardial infarction or abnormal creatinine
* History of known food allergy and/or dietary restriction
* Diabetes requiring insulin
* Pregnancy
* Diarrhea defined as watery stools more than 3 times a day for more than 3 days

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Fasting insulin | 4 weeks

SECONDARY OUTCOMES:
Gene Expression | One month

CONTACTS AND LOCATIONS:
Overall Officials: Simin Liu, M.D., Sc.D, Principal Investigator — UCLA Program on Genomics and Nutrition; James Sul, M.D., Principal Investigator — UCLA Program on Genomics and Nutrition
Locations (1):
- UCLA General Clinical Research Center, Los Angeles, California, United States

REFERENCES:
- [Result] Chacko SA, Sul J, Song Y, Li X, LeBlanc J, You Y, Butch A, Liu S. Magnesium supplementation, metabolic and inflammatory markers, and global genomic and proteomic profiling: a randomized, double-blind, controlled, crossover trial in overweight individuals. Am J Clin Nutr. 2011 Feb;93(2):463-73. doi: 10.3945/ajcn.110.002949. Epub 2010 Dec 15. PMID 21159786